CLINICAL TRIAL: NCT00198263
Title: An Open-Label Study Using the Medpulser® Electroporation System to Treat Head and Neck Cancer
Brief Title: Study Using the Medpulser Electroporation System With Bleomycin to Treat Head and Neck Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-HNBE-2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; cancer; bleomycin; medpulser; electroporation; primary oral cavity, primary pharyngeal, primary laryngeal, salivary gland, limited recurrent and second primary tumors
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Bleomycin

STUDY DESIGN:
Intervention Model Description: Medpulser electroporation with Bleomycin
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bleomycin (Experimental): Bleomycin 4 USP Units/mL; intratumorally at dose of 0.25mL/cm^3
  Interventions: Combination Product: Medpulser Electroporation with Bleomycin

INTERVENTIONS:
Combination Product: Medpulser Electroporation with Bleomycin — The MedPulser device will be used in conjunction with injection of Bleomycin Sulfate at a concentration of 1 U/ml per cm3 of tumor treatment area.

SUMMARY:
The purpose of the trial is to study the safety and efficacy of the Medpulser Electroporation System with bleomycin in the treatment of head and neck cancer.

DETAILED DESCRIPTION:
Electroporation therapy is a tumor-specific ablative treatment modality with the potential to manage local tumors without the potentially undesirable side effects of systemic chemotherapy agents or radiotherapy. Surgical resection of solid tumors often leaves subjects with significant organ dysfunction and/or permanent disfigurement requiring reconstructive surgery. In contrast, electroporation therapy may offer equivalent disease control to conventional surgery with lessened need for reconstructive surgery. Electroporation therapy may also provide economic benefits over conventional surgical and or radiation procedures through reduced operating theatre costs, hospital stays and post treatment interventions. The ability to shrink or eliminate local tumors with the MedPulser® System when used in conjunction with intralesional Bleomycin is an important new possible treatment for the conservative local management of SCCHN and provides a possible alternative treatment option to surgical excision in the management of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of primary oral cavity, primary pharyngeal, primary laryngeal, salivary gland, limited recurrent and second primary tumors must be confirmed by histological examination of a tissue sample (e.g., biopsy) obtained within 2 months of the subject receiving the study treatment.
2. The length of the longest diameter of the study lesion must be < 5 cm and the calculated treatment volume (tumor volume plus a 0.5 cm margin around the tumor) for the study lesion [where treatment volume = 0.5 (a+1) (b+1)2 and where a = length of the longest diameter (cm), b = the next longest diameter perpendicular to "a" (cm)] must be < 60.0 cm3.
3. Age: 18 years or older.
4. Male or female.
5. Men and women of childbearing potential must be using Investigator prescribed contraceptive methods while undergoing protocol related therapy.
6. Baseline performance status: ECOG 0-2:

   * Grade 0: Fully active, able to carry on all pre-disease performance without restriction.
   * Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
   * Grade 2: Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
7. Life expectancy of at least 6 months.
8. Subjects must sign a written Informed Consent prior to receiving any study procedures or treatments.

Exclusion Criteria:

1. Subjects with tumors suspected of involving a 50% or greater encasement of a blood vessel as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
2. Subjects with tumors having bone invasion.
3. Subjects with hypersensitivity to bleomycin.
4. Subjects who have received or will exceed a total lifetime dose of bleomycin greater than 400 units.
5. Subjects deemed unsuitable for general anesthesia.
6. Subjects with a significant history of emphysema or pulmonary fibrosis.
7. Subjects with indwelling cardiac pacemakers who cannot tolerate a period with pacemaker turned off.
8. Subjects with a history of uncontrolled cardiac arrhythmia.
9. Women who are pregnant, or are nursing. Women must have a negative pregnancy test (urine pregnancy tests are acceptable) within 7 days of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2004-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To characterize local tumor recurrence through 8 months post-EPT/bleomycin treatment | 8 Months

SECONDARY OUTCOMES:
To measure pharmacoeconomic factors (hospital costs, extent of medical interventions, medication use) in subjects treated by EPT/bleomycin | 24 Months
To evaluate organ function and appearance using the Performance Status Scale (PSS) and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck (EORTC QLQ - H&N 35) at 4 and 8 months following treatment | 4 and 8 Months
To document the performance of the MedPulser® System during EPT/bleomycin treatment | 8 Nonths
To monitor local and systemic adverse events through the Month 4 follow-up study visit | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goldfarb, MD, Study Chair — Inovio Pharmaceuticals
Locations (1):
- Inovio Biomedical Corporation, San Diego, California, United States